CLINICAL TRIAL: NCT00005964
Title: Randomized Phase II Study of Dose-Adjusted EPOCH vs. NHL-15 Chemotherapy for Patients With Previously Untreated Aggressive Non-Hodgkin's Lymphoma (NHL)
Brief Title: Comparison of Two Combination Chemotherapy Regimens in Treating Patients With Previously Untreated Aggressive Stage II, Stage III, or Stage IV Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-C59910; U10CA031946 (NIH); CLB-C59910; CDR0000067947 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-07-05; First posted 2003-11-05 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy + prednisone + filgrastim (Experimental): Patients receive doxorubicin IV, etoposide IV, vincristine IV, and cyclophosphamide IV continuously over days 1-4. Patients also receive oral prednisone twice daily on days 1-5 and filgrastim (G-CSF) subcutaneously beginning on day 6 until blood counts recover. Treatment continues every 21 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective in treating aggressive non-Hodgkin's lymphoma.

PURPOSE: Randomized phase II trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have previously untreated aggressive stage II, stage III, or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rates in patients with previously untreated aggressive non-Hodgkin's lymphoma treated with doxorubicin, etoposide, vincristine, cyclophosphamide, and prednisone (EPOCH). II. Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive doxorubicin IV, etoposide IV, vincristine IV, and cyclophosphamide IV continuously over days 1-4. Patients also receive oral prednisone twice daily on days 1-5 and filgrastim (G-CSF) subcutaneously beginning on day 6 until blood counts recover. Treatment continues every 21 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage II, III, or IV non-Hodgkin's lymphoma (NHL) Diffuse large B-cell lymphoma (including immunoblastic features) OR Anaplastic large cell lymphoma No mantle cell lymphomas including equivocal B-cell lymphomas that are CD5+ and CD23-, have t(11;14), or express markers of mantle cell lymphoma or other subtypes No low-grade lymphoma (e.g., follicular center cells in bone marrow) Patients who have 3-5 International Prognostic Index risk factors must have refused participation in SWOG-S9704/CALGB-59903 trial No known lymphomatous CNS involvement, including parenchymal or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: Not specified Performance status: 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3* Platelet count at least 100,000/mm3* *unless attributable to NHL Hepatic: Bilirubin no greater than 2.0 mg/dL (without Gilbert's disease)* *unless attributable to NHL Renal: Creatinine no greater than 1.5 mg/dL* *unless attributable to NHL Cardiovascular: LVEF greater than 45% No ischemic heart disease No myocardial infarction or congestive heart failure in past year Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cytotoxic chemotherapy No other concurrent chemotherapy Endocrine therapy: Prior glucocorticoids allowed (less than 10 day course) for urgent local disease at diagnosis (e.g., cord compression, superior vena cava syndrome) No concurrent dexamethasone (except as indicated by protocol) or other steroidal antiemetics No concurrent hormonal therapy except for non-disease related conditions Radiotherapy: Prior limited field radiotherapy allowed Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2000-05; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zelenetz, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (47):
- United States (47):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia